CLINICAL TRIAL: NCT05148455
Title: Total Body Dermoscopic Evaluation of Pregnancy-related Changes in Melanocytic Nevi Using the FotoFinder ATBM Master System and the Impact of Artificial Intelligence Assisted Examinations on the Patients' Skin Cancer Screening Experience: A Prospective Two-arm Controlled Observational Study
Brief Title: Pregnancy-related Changes in Melanocytic Nevi
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02494; th21Maul2
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Melanocytic Nevi (MN)
Keywords: skin cancer screening; total body mapping; deep learning-driven body scan; FotoFinder® ATBM master; malignant melanoma; pregnancy-related changes in melanocytic nevi
MeSH Terms: conditions — Nevus, Pigmented; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women
  Interventions: Other: standard-of-care clinical skin examination; Diagnostic Test: skin assessment with the 2D FotoFinder ATBM master system; Other: data collection by participant questionnaire
- non-pregnant women (control group)
  Interventions: Other: standard-of-care clinical skin examination; Diagnostic Test: skin assessment with the 2D FotoFinder ATBM master system; Other: data collection by participant questionnaire

INTERVENTIONS:
Other: standard-of-care clinical skin examination — inspection of melanocytic nevi by dermatologist
Diagnostic Test: skin assessment with the 2D FotoFinder ATBM master system — The FotoFinder® ATBM master device provides the combination of total body mapping with deep learning-driven body scan algorithm which identifies all pigmented skin lesions of the body surface by pattern recognition software and supplies a risk assessment score (0.0-1.0; 0 indicating no suspicion for melanoma, 1 indicating a high suspicion for melanoma).The integrated software analyzer scores regarding malignancy probability of the moles (FotoFinder® score: 0.0-1.0) will be collected.
Other: data collection by participant questionnaire — At baseline, the participants will complete a questionnaire concerning their previous exposure to sun, their current sun-related protective behaviours, their history of skin check frequency and skin cancer at baseline. Additionally, in each consultation newly-created study-specific questions concerning the participants' examination experience, the sun-related protective behaviours and worries about skin cancer throughout the study will be investigated.

SUMMARY:
This study is

* to analyze whether more changes in melanocytic nevi (MN) occur in women during and after pregnancy compared to non-pregnant women of the same age
* and to analyze psychological effects of total body mapping and dermoscopic examination assisted by artificial intelligence during pregnancy.

DETAILED DESCRIPTION:
Melanocytic nevi (MN) are believed to undergo macroscopic and dermoscopic alterations during pregnancy. Possible changing features previously observed include color, pigment network, size, vascularization and the emerging of dots and globules. Recent studies have reported of melanoma being associated with increased mortality in pregnant women when compared to non-pregnant women. The new FotoFinder® ATBM master device provides the combination of total body mapping with deep learning-driven body scan algorithm which identifies all pigmented skin lesions of the body surface by pattern recognition software and supplies a risk assessment score (0.0-1.0; 0 indicating no suspicion for melanoma, 1 indicating a high suspicion for melanoma).

This study is

* to analyze whether more changes in melanocytic nevi (MN) occur in women during and after pregnancy compared to non-pregnant women of the same age
* and to analyze psychological effects of total body mapping and dermoscopic examination assisted by artificial intelligence during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female participants beyond the 12th week of pregnancy
* Non-pregnant female participants

Exclusion Criteria:

* Fitzpatrick skin phototypes V and VI
* less than 15 MN (MN with a diameter less than 2mm will not be taken into account)
* insufficient knowledge of project language (German, English, French)
* inability to give consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant volunteers recruited through the Department of Gynaecology and Obstetrics at the University Hospital of Basel and through study advertisement displayed at gynaecological practices in the city of Basel.
  Non-pregnant volunteers recruited through study advertisement displayed at the University of Basel and at the Department of Dermatology at the University Hospital Basel and through an advertisement.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Change in macroscopic aspect of melanocytic nevi | for pregnant women: Visit 1 (between the 12th and 16th week of pregnancy), Visit 2 (between the 29th and 33rd week of pregnancy), Visit 3 (between 8 to 12 weeks after delivery). Non- pregnant women: Visit 1, Visit 2 (17 to 21 weeks after Visit 1)
  Change in macroscopic aspect of melanocytic nevi
Change in mole analyzer score with the 2D FotoFinder ATBM master system | for pregnant women: Visit 1 (between the 12th and 16th week of pregnancy), Visit 2 (between the 29th and 33rd week of pregnancy), Visit 3 (between 8 to 12 weeks after delivery). Non- pregnant women: Visit 1, Visit 2 (17 to 21 weeks after Visit 1)
  mole analyzer score (0.0-1.0; 0 indicating no suspicion for melanoma, 1 indicating a high suspicion for melanoma)

SECONDARY OUTCOMES:
Change in number of new malignant melanoma | for pregnant women: Visit 1 (between the 12th and 16th week of pregnancy), Visit 2 (between the 29th and 33rd week of pregnancy), Visit 3 (between 8 to 12 weeks after delivery). Non- pregnant women: Visit 1, Visit 2 (17 to 21 weeks after Visit 1)
  Change in number of new malignant melanoma
Change in psychological impact of skin cancer screening by descriptive analyzes of participants questionnaire | for pregnant women: Visit 1 (between the 12th and 16th week of pregnancy), Visit 2 (between the 29th and 33rd week of pregnancy), Visit 3 (between 8 to 12 weeks after delivery). Non- pregnant women: Visit 1, Visit 2 (17 to 21 weeks after Visit 1)
  Change in psychological impact of skin cancer screening by descriptive analyzes of participants questionnaire (investigating the subjective examination experience, the impact on skin cancer worries and the participants' sun protection and self-inspection behaviour).

CONTACTS AND LOCATIONS:
Overall Officials: Lara Valeska Maul, Dr. med., Principal Investigator — University Hospital Basel, Department of Dermatology
Locations (1):
- University Hospital Basel, Department of Dermatology, Basel, Switzerland